CLINICAL TRIAL: NCT03496064
Title: Bernese-European RegistrY for Ischemic Stroke Patients Treated Outside Current Guidelines With Neurothrombectomy Devices Using the SOLITAIRE™ FR With the Intention For Thrombectomy
Brief Title: Registry for Evaluating Outcome of Acute Ischemic Stroke Patients Treated With Mechanical Thrombectomy.
Acronym: BEYOND-SWIFT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Toulouse (Other); Technical University of Munich (Other); University of Toronto (Other); Medtronic (Industry); CHU de Reims (Other); Hospital Vall d'Hebron (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 231/2014
Record Dates: First submitted 2018-03-27; First posted 2018-04-12 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Stroke
Keywords: Thrombectomy; Eligibility; Large vessel occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (6):
- Anterior circulation LVO patients with ASPECTS <6
  Interventions: Other: Successful reperfusion
- Anterior circulation LVO patients with NIHSS<8
- Posterior versus anterior circulation LVO patients
- LVO patients with isolated PCA or ACA occlusions
  Interventions: Other: Successful reperfusion
- Tandem lesions versus non-tandem lesion
- Bridging vs Direct MT

INTERVENTIONS:
Other: Successful reperfusion — Defined as modified Thrombolysis in Cerebral Infarction 2b/3
  Groups: Anterior circulation LVO patients with ASPECTS <6; LVO patients with isolated PCA or ACA occlusions

SUMMARY:
The Bernese-European RegistrY for ischemic stroke patients treated Outside current guidelines with Neurothrombectomy Devices using the SOLITAIRE™ FR With the Intention For Thrombectomy (BEYOND-SWIFT) is a retrospective, multi-center, non-randomized observational study aims to investigate the safety and efficacy of a Medtronic market-released neurothrombectomy device (applied as initial devices used for intervention) in acute ischemic stroke patients who do not fulfill treatment eligibility according to current guidelines. Patients will be treated or were treated at the discretion of the investigator, independent of participation in this registry. Primary Analysis is the Impact of successful reperfusion on functional outcome at day 90 in patients presenting with large infarct cores (ASPECTS<6) or minor symptoms (NIHSS<8).

ELIGIBILITY:
Inclusion Criteria:

* Patients or patient's legally authorized representative have given informed consent according to Good Clinical Practices (GCP) and/or IRB and/or local or institutional policies.
* The patient presents with an intracranial large vessel occlusion and therewith-related neurological symptoms and has been or will be treated with a Medtronic marketed-release neurothrombectomy device (applied as first device to attempt retrieving the thrombus).

Exclusion Criteria:

* Current participation in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with large-vessel occlusion acute ischemic stroke subjected to endovascular treatment using a Medtronic market-released neurothrombectomy device (applied as initial devices used for intervention).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
3 month functional independence | 0-90 days
  Number of patients with modified Rankin Scale <=2
Favourable outcome | 0-90 days
  Number of patients with modified Rankin Scale <=3
Excellent outcome | 0-90 days
  Number of patients with modified Rankin Scale <=1

SECONDARY OUTCOMES:
Successful reperfusion | Day 0
  Number of patients with modified Thrombolysis in Cerebral Infarction 2b / 3
Symptomatic intracranial hemorrhage | Day 0-1
  Number of patients with symptomatic intracranial hemorrhage according to ECASSII definition
Time to reperfusion | Day 0
  Groin puncture to TICI2b/3
Mortality | Day 0-90
  Number of patients with modified Rankin Scale 6

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, MD, MSc, Principal Investigator — Department of Neurology, University Hospital Bern, Switzerland; Jan Gralla, MD, Principal Investigator — Department of Neuroradiology, University Hospital Bern, Switzerland
Locations (1):
- Dept. of Neurology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mujanovic A, Kurmann CC, Dobrocky T, Olive-Gadea M, Maegerlein C, Pierot L, Mendes Pereira V, Costalat V, Psychogios M, Michel P, Beyeler M, Piechowiak EI, Seiffge DJ, Mordasini P, Arnold M, Gralla J, Fischer U, Kaesmacher J, Meinel TR; BEYOND-SWIFT Investigators. Bridging intravenous thrombolysis in patients with atrial fibrillation. Front Neurol. 2022 Aug 3;13:945338. doi: 10.3389/fneur.2022.945338. eCollection 2022. PMID 35989924
- [Derived] Kaesmacher J, Maamari B, Meinel TR, Piechowiak EI, Mosimann PJ, Mordasini P, Goeldlin M, Arnold M, Dobrocky T, Boeckh-Behrens T, Berndt M, Michel P, Requena M, Benali A, Pierot L, Mendes Pereira V, Boulouis G, Brehm A, Sporns PB, Ospel JM, Gralla J, Fischer U; BEYOND-SWIFT Investigators. Effect of Pre- and In-Hospital Delay on Reperfusion in Acute Ischemic Stroke Mechanical Thrombectomy. Stroke. 2020 Oct;51(10):2934-2942. doi: 10.1161/STROKEAHA.120.030208. Epub 2020 Sep 16. PMID 32933420
- [Derived] Meinel TR, Kaesmacher J, Mosimann PJ, Seiffge D, Jung S, Mordasini P, Arnold M, Goeldlin M, Hajdu SD, Olive-Gadea M, Maegerlein C, Costalat V, Pierot L, Schaafsma JD, Fischer U, Gralla J. Association of initial imaging modality and futile recanalization after thrombectomy. Neurology. 2020 Oct 27;95(17):e2331-e2342. doi: 10.1212/WNL.0000000000010614. Epub 2020 Aug 26. PMID 32847948
- [Derived] Meinel TR, Kniepert JU, Seiffge DJ, Gralla J, Jung S, Auer E, Frey S, Goeldlin M, Mordasini P, Mosimann PJ, Nogueira RG, Haussen DC, Rodrigues GM, Uphaus T, L'Allinec V, Krajickova D, Alonso A, Costalat V, Hajdu SD, Olive-Gadea M, Maegerlein C, Pierot L, Schaafsma J, Suzuki K, Arnold M, Heldner MR, Fischer U, Kaesmacher J. Endovascular Stroke Treatment and Risk of Intracranial Hemorrhage in Anticoagulated Patients. Stroke. 2020 Mar;51(3):892-898. doi: 10.1161/STROKEAHA.119.026606. Epub 2020 Jan 29. PMID 31992179
- [Derived] Meinel TR, Kaesmacher J, Mordasini P, Mosimann PJ, Jung S, Arnold M, Heldner MR, Michel P, Hajdu SD, Ribo M, Requena M, Maegerlein C, Friedrich B, Costalat V, Benali A, Pierot L, Gawlitza M, Schaafsma J, Pereira VM, Gralla J, Fischer U. Outcome, efficacy and safety of endovascular thrombectomy in ischaemic stroke according to time to reperfusion: data from a multicentre registry. Ther Adv Neurol Disord. 2019 Mar 27;12:1756286419835708. doi: 10.1177/1756286419835708. eCollection 2019. PMID 30944585
- [Derived] Kaesmacher J, Chaloulos-Iakovidis P, Panos L, Mordasini P, Michel P, Hajdu SD, Ribo M, Requena M, Maegerlein C, Friedrich B, Costalat V, Benali A, Pierot L, Gawlitza M, Schaafsma J, Mendes Pereira V, Gralla J, Fischer U. Mechanical Thrombectomy in Ischemic Stroke Patients With Alberta Stroke Program Early Computed Tomography Score 0-5. Stroke. 2019 Apr;50(4):880-888. doi: 10.1161/STROKEAHA.118.023465. PMID 30827193

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03496064/SAP_000.pdf